CLINICAL TRIAL: NCT00017602
Title: Randomized Phase III Study of Dexamethasone With or Without Genasense (Bcl-2 Antisense Oligonucleotide) in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Dexamethasone With or Without Oblimersen in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genta Incorporated (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068722; GENTA-GMY302; UF-G-29-2001
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2003-08

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — oblimersen; Dexamethasone

INTERVENTIONS:
Biological: oblimersen sodium
Drug: dexamethasone

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Oblimersen may increase the effectiveness of dexamethasone by making cancer cells more sensitive to the drug. It is not yet known if dexamethasone is more effective with or without oblimersen in treating multiple myeloma.

PURPOSE: Randomized phase III trial to compare the effectiveness of dexamethasone with or without oblimersen in treating patients who have relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the time to disease progression in patients with relapsed or refractory multiple myeloma treated with dexamethasone with or without oblimersen.
* Compare the duration of response and objective response rate in patients treated with these regimens.
* Compare the proportion of patients without disease progression after 6 months and the proportion of patients who have not discontinued treatment after 6 months in these two patient groups.
* Compare the safety of these regimens in these patients.
* Compare survival of patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to response to prior therapy (relapsed vs refractory), prior autologous stem cell transplantation (yes vs no), and number of prior therapy regimens (1-2 vs 3-6). Patients are randomized to 1 of 2 treatment arms.

Arm I

* Induction: Patients receive oblimersen (G3139) IV continuously on days 1-7 and 15-21 and oral dexamethasone daily on days 4-7, 11-14, and 18-21.
* Maintenance: One week after completion of induction therapy, patients with stable or responsive disease receive G3139 IV continuously on days 1-7 and oral dexamethasone daily on days 4-7. Courses repeat every 3 weeks for a maximum of 1 year in the absence of disease progression or unacceptable toxicity.

Arm II

* Induction: Patients receive oral dexamethasone daily for 4 days on weeks 1-3.
* Maintenance: One week after completion of induction therapy, patients with stable or responsive disease receive oral dexamethasone daily for 4 days. Courses repeat every 3 weeks for a maximum of 1 year in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 months for 2 years.

PROJECTED ACCRUAL: A total of 200 patients (100 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: NOTE: This trial is being conducted at many institutions throughout the country. Please contact Genta for a site near you.

* Progressive multiple myeloma defined by one of the following:

  * Primary resistance or progressive disease after achieving less than a partial response after at least 2 courses of combination chemotherapy (that included at least 1 myelosuppressive drug) within the past 3 months
  * Relapsed or progressive disease after at least a partial response to prior therapy
  * Progressive disease after high-dose chemotherapy and autologous stem cell transplantation
* Progressive disease defined by at least 1 of the following:

  * Increase in serum M-protein by at least 50% or at least 2 g/dL above the lowest remission or baseline level
  * Increase in urinary M-protein by at least 50% or at least 2 g/24 hours above lowest remission or baseline level
  * Appearance of new lytic bone lesions or at least 50% increase in size of an existing bone lesion
* Quantifiable serum and/or urine paraprotein
* Bone marrow plasmacytosis at least 5% of total nucleated cells
* Measurable disease

  * Serum M-protein level at least 1.0 g/dL OR
  * Urinary M-protein excretion at least 200 mg/24 hours

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-3

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,000/mm3
* Platelet count at least 50,000/mm3
* No bleeding or coagulation disorder

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST no greater than 2.5 times ULN
* PT and PTT no greater than 1.5 times ULN
* No history of chronic hepatitis or cirrhosis

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No active symptoms of coronary artery disease (e.g., uncontrolled arrhythmias or recurrent chest pain despite prophylactic medication)
* No New York Heart Association class III or IV heart disease
* No uncontrolled congestive heart failure
* No grade 2 or greater cardiovascular signs or symptoms within the past 4 weeks

Other:

* HIV negative
* No active peptic ulcer disease
* No uncontrolled seizure disorder
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No active uncontrolled infection
* No active autoimmune disease
* No hypersensitivity to phosphorothioate-containing oligonucleotides or to dexamethasone
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* At least 3 weeks since prior immunotherapy
* At least 72 hours since prior thalidomide
* Concurrent epoetin alfa allowed

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosourea)

Endocrine therapy:

* At least 3 weeks since prior corticosteroids
* No concurrent chronic corticosteroids

Radiotherapy:

* At least 14 days since prior radiotherapy except limited radiotherapy to a single bone lesion

Surgery:

* At least 3 weeks since prior major surgery
* No prior organ allograft

Other:

* At least 4 weeks since other prior investigational therapy
* No more than 6 prior therapies for myeloma
* No concurrent immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-12; Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley R. Frankel, MD, Study Chair — Genta Incorporated
Locations (1):
- Genta Incorporated, Berkeley Heights, New Jersey, United States

REFERENCES:
- [Result] Chanan-Khan AA, Niesvizky R, Hohl RJ, Zimmerman TM, Christiansen NP, Schiller GJ, Callander N, Lister J, Oken M, Jagannath S. Phase III randomised study of dexamethasone with or without oblimersen sodium for patients with advanced multiple myeloma. Leuk Lymphoma. 2009 Apr;50(4):559-65. doi: 10.1080/10428190902748971. PMID 19373653